CLINICAL TRIAL: NCT05010603
Title: Late Onset Alzheimer's Disease
Acronym: LOAD
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAAP0479; 5U24AG056270 (NIH)
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease
Keywords: Genetic testing; Genetic influence
MeSH Terms: conditions — Alzheimer Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and samples from autopsy/brain tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Families with a history of Alzheimer's Disease: Families with two or more family members affected with Alzheimer's Disease
  Interventions: Genetic: Blood Draw; Other: Late Onset Alzheimer's Disease (LOAD) Neuropsychological Battery Test
- Un-related, non-demented controls: Un-related, non-demented healthy controls over age 55
  Interventions: Genetic: Blood Draw; Other: Late Onset Alzheimer's Disease (LOAD) Neuropsychological Battery Test
- Individuals with Dementia (Alzheimer's Disease): Individuals with dementia over the age of 65
  Interventions: Genetic: Blood Draw; Other: Late Onset Alzheimer's Disease (LOAD) Neuropsychological Battery Test

INTERVENTIONS:
Genetic: Blood Draw — Collection of blood samples for genetic testing
Other: Late Onset Alzheimer's Disease (LOAD) Neuropsychological Battery Test — Memory Test

SUMMARY:
The goal of this study is to is to focus on the genetic influences on Alzheimer's Disease (AD) risk. The investigators are looking for families and/or individuals (affected or unaffected) of any ethic background (African American, Caucasian, and Hispanics) with a family history of AD and willing to participate.

DETAILED DESCRIPTION:
The purpose of this study is to focus on the genetic influences on Alzheimer's disease (AD) risk. Specifically, the investigators hypothesize that one or more genes, other than the previously identified susceptibility gene apolipoprotein-E (APOE), or the 3 genes associated with early-onset familial AD, presenilin-1 (PS-1), presenilin-2 (PS-2) or B-amyloid precursor protein (APP), increase the risk of AD in families with multiple individuals affected with AD. The investigators propose to test this hypothesis by performing genetic linkage analysis in order to detect the chromosomal location of genes that may increase the risk of Alzheimer's disease. In addition, the investigators will study genes known to increase the risk of Alzheimer's disease and other related disorders such as early onset AD, Pick disease, corticobasal degeneration, progressive supranuclear palsy, and familial frontotemporal dementia with parkinsonism and Lewy Body Dementia.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of definite or probable AD or have a diagnosis of a related neurodegenerative disorder such as Frontotemporal Dementia (FTD) or Lewy Body Dementia (LBD) (will also recruit sporadic FTD and LBD) cases.
* a living sibling with probable or possible AD;
* a third living relative affected with AD (onset age 50 or older) or unaffected (60 or older);
* participants in the proband's generation with an identified companion serving as an informant;
* participants who have capacity to consent or participants lacking capacity to consent with a surrogate/proxy in place to provide consent.

Exclusion Criteria:

* failure to identify an appropriate informant;
* uncertainty of the clinical diagnosis of Alzheimer's disease or other related disorder;
* discovery of additional diagnosis that could account for the clinical manifestations;
* unwillingness to participate;
* failure to identify a living sibling with AD or other related disorder (except in the cases of sporadic FTD and sporadic LBD);
* participants lacking the capacity to consent who do not have a surrogate or proxy or next of kin to provide consent.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators intend to recruit individuals from: 1) community-based studies; 2) the Alzheimer's Disease Research Center Memory Disorders Center; 3) the private offices of the study neurologists; 4) public recruitment; 5) referrals from the Alzheimer's Association; 6) referrals from the NCRAD; 7)previously unidentified members of existing families not previously recruited. The investigators will also use advertisements such as radio, television and newspapers.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-11-15 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Total number of genes identified to be associated with the risk of AD | 5 years
  Genetic Linkage Analysis to Identify Genes Associated with the risk of Alzheimer's Disease: Identification of genes by performing genetic linkage analysis, in order to detect the chromosomal location of genes that may increase the risk of Alzheimer's disease.

CONTACTS AND LOCATIONS:
Overall Officials: Richard P. Mayeux, MD, MSc, Principal Investigator — Columbia University
Locations (12):
- United States (12):
  - University of Washington, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Rush University, Aurora, Illinois
  - Indiana University, Bloomington, Indiana
  - NCRAD at Indiana University, Indianapolis, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Joanne Norton, St Louis, Missouri
  - Columbia University Irving Medical Center, New York, New York
  - North Carolina State University, Raleigh, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data is stored in a secured database at Columbia University and de-identified data will be sent to the National Cell Repository for Alzheimer's disease. DNA will be stored at the National Cell Repository for Alzheimer's disease (NCRAD) at Indiana University. In addition to the blood sample, year of birth, family history of dementia, and diagnosis will be sent to NCRAD. DNA and associated clinical and demographic data will be made available to qualified and approved researchers studying the genetics of AD, aging, and related disorders. If the participant agrees, his/her de-identified samples and data will be made available to investigators studying the genetics of any human disease. Identity of participants will not be shared with NCRAD or with any investigators.
Supporting Information: Study Protocol
Time Frame: The data is currently available
Access Criteria: When requesting samples to NCRAD the "Master Agreement for Transfer of Materials to NCRAD" and related Appendix A must be completed prior to the transfer of any samples. The Master Material Transfer Agreement (MTA) agreement is between the Institutions and is not Investigator specific. Therefore, if you think your Institution may already have a Master MTA in place with NCRAD.
URL: https://osp.od.nih.gov